CLINICAL TRIAL: NCT04976270
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Oral Doses of GLPG3667 in Adult, Healthy Male Subjects
Brief Title: A Study to Evaluate How Well Single and Multiple Doses of GLPG3667 Are Tolerated in Healthy, Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GLPG3667-CL-118; 2021-002488-23 (EudraCT Number)
Record Dates: First submitted 2021-07-19; First posted 2021-07-26 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GLPG3667 SD (Experimental): Participants will receive a single dose of GLPG3667
  Interventions: Drug: GLPG3667
- Placebo SD (Placebo Comparator): Participants will receive a single dose of matching placebo
  Interventions: Drug: Placebo
- GLPG3667 MD (Experimental): Participants will receive repeated doses of GLPG3667 for 13 days.
  Interventions: Drug: GLPG3667
- Placebo MD (Placebo Comparator): Participants will receive repeated doses of matching placebo for 13 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG3667 — GLPG3667 capsules
  Arms: GLPG3667 MD; GLPG3667 SD
Drug: Placebo — Matching placebo capsules
  Arms: Placebo MD; Placebo SD

SUMMARY:
This study is a phase I, randomized, double-blind, placebo-controlled, single-center, to evaluate the safety, tolerability, and pharmacokinetics (PK) of GLPG3667 after an oral single dose (SD) of GLPG3667 (part 1) and after oral multiple doses (MD) for 13 days of GLPG3667 (part 2) in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male between 18 and 55 years of age (extremes included), on the date of signing the informed consent form (ICF).
* A body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive.
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and fasting clinical laboratory safety tests, available at screening and prior to randomization. Hemoglobin, neutrophil, lymphocyte, and platelet counts must be above the lower limit of normal range. Total bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) must be below the upper limit of normal. Other clinical laboratory safety test results must be within the reference ranges or test results that are outside the reference ranges need to be considered not clinically significant in the opinion of the investigator.

This list only contains the key inclusion criteria.

Exclusion Criteria:

* Known hypersensitivity to investigational product (IP) ingredients or history of a significant allergic reaction to IP ingredients as determined by the investigator.
* Positive serology for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) or history of hepatitis from any cause with the exception of hepatitis A that has resolved at least 3 months prior to first dosing of the IP.

This list only contains the key exclusion criteria.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events, and TEAEs leading to treatment discontinuations | From screening through study completion, an average of 3 months
  To evaluate the safety and tolerability of single and multiple oral doses of GLPG3667, in adult, healthy, male subjects compared with placebo

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of GLPG3667 - SD | Between Day 1 pre-dose and Day 4
  To evaluate the PK of single and multiple oral doses of GLPG3667 in adult, healthy male subjects.
Maximum observed plasma concentration (Cmax) of GLPG3667 - MD | Between Day 1 pre-dose and Day 16
  To evaluate the PK of single and multiple oral doses of GLPG3667 in adult, healthy male subjects.
Area under the plasma concentration-time curve (AUC) of GLPG3667 - SD | Between Day 1 pre-dose and Day 4
  To evaluate the PK of single and multiple oral doses of GLPG3667 in adult, healthy male subjects.
Area under the plasma concentration-time curve (AUC) of GLPG3667 - MD | Between Day 1 pre-dose and Day 16
  To evaluate the PK of single and multiple oral doses of GLPG3667 in adult, healthy male subjects.
Terminal elimination half-life (t1/2) of GLPG3667 - SD | Between Day 1 pre-dose and Day 4
  To evaluate the PK of single and multiple oral doses of GLPG3667 in adult, healthy male subjects.
Terminal elimination half-life (t1/2) of GLPG3667 - MD | Between Day 1 pre-dose and Day 16
  To evaluate the PK of single and multiple oral doses of GLPG3667 in adult, healthy male subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Rueda-Rincon, MD, PhD, Study Director — Galapagos NV
Locations (1):
- Drug Research Unit Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No